CLINICAL TRIAL: NCT01726036
Title: Gomco Versus Mogen: Which is Best? A Randomized Controlled Trial: The GMRT Study.
Brief Title: Gomco Versus Mogen: Which is Best? A Randomized Controlled Trial
Acronym: GMRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-11121
Record Dates: First submitted 2012-11-01; First posted 2012-11-14 (Estimated); Results first posted 2019-05-16 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-01

CONDITIONS: Circumcision, Male
Keywords: neonatal circumcision; neonatal surgical pain; Mogen; Gomco

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gomco Circumcision Clamp (Active Comparator): Gomco circumcision clamp used for neonatal circumcision.
  Interventions: Device: Gomco Circumcision Clamp
- Mogen Circumcision Clamp (Active Comparator): Mogen circumcision clamp used for neonatal circumcision.
  Interventions: Device: Mogen Circumcision Clamp

INTERVENTIONS:
Device: Gomco Circumcision Clamp — Neonatal male circumcision utilizing the Gomco Circumcision Clamp
  Arms: Gomco Circumcision Clamp
Device: Mogen Circumcision Clamp — Neonatal male circumcision utilizing the Mogen Circumcision Clamp
  Arms: Mogen Circumcision Clamp

SUMMARY:
The purpose of this study is to compare two commonly used circumcision clamps (Gomco and Mogen) to see which results in less neonatal pain.

DETAILED DESCRIPTION:
Objective: To compare pain levels assessed by salivary cortisol and standardized neonatal pain scale among the two most common infant circumcision techniques in uncomplicated pregnancies after a thorough resident-wide education curriculum under attending physician supervision.

The secondary objectives are to assess the operative time, complication rates such as infection and bleeding and short term outcomes including need for re-circumcision among treatment groups.

Hypothesis: The Mogen technique of circumcision is less painful, faster, and associated with less bleeding for newborns when compared to the Gomco technique after a resident circumcision standard teaching curriculum.

ELIGIBILITY:
Inclusion Criteria:

* term infants delivered by cesarean section or vaginal delivery at Good Samaritan Hospital during the time period of the study
* Infants with no blood drawn two hours prior to the circumcision
* Singletons

Exclusion Criteria:

* Infants with congenital anomalies and/or known chromosomal syndromes
* Preterm infants defined as less than 37 / 0 weeks gestation.
* Delivery secondary to non-reassuring fetal heart tracing, defined by the delivering physician
* Infants of diabetic mothers.
* Infants of preeclamptic mothers on magnesium sulfate within 48 hours of delivery.
* Infants delivered by vacuum-assisted or forceps-assisted vaginal delivery.
* Infants of mothers who took steroids for fetal lung maturity within 7 days of delivery. (This may apply to term infants if the mother had no prenatal care and her gestational age was not known on arrival).
* Infants with a 5 minutes apgar score of less than 7
* Infants born to mothers with a history of drug abuse during pregnancy, currently on methadone, or with Hepatitis C or HIV.

Max Age: 4 Days | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mounira Habli, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared by manuscript.

REFERENCES:
- [Derived] Sinkey RG, Eschenbacher MA, Walsh PM, Doerger RG, Lambers DS, Sibai BM, Habli MA. The GoMo study: a randomized clinical trial assessing neonatal pain with Gomco vs Mogen clamp circumcision. Am J Obstet Gynecol. 2015 May;212(5):664.e1-8. doi: 10.1016/j.ajog.2015.03.029. Epub 2015 Mar 17. PMID 25794628

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 274 infants were enrolled into the study from 10/2012 through 6/2013.
Groups:
- Gomco Circumcision Clamp: Gomco circumcision clamp used for neonatal circumcision.
  Gomco Circumcision Clamp
- Mogen Circumcision Clamp: Mogen circumcision clamp used for neonatal circumcision.
  Mogen Circumcision Clamp
Period: Overall Study
Arm/Group | Gomco Circumcision Clamp | Mogen Circumcision Clamp
Started | 137 | 137
Completed | 121 | 130
Not Completed | 16 | 7

BASELINE CHARACTERISTICS:
Population: Male infants receiving circumcisions
Groups:
- Total: Total of all reporting groups
Arm/Group | Gomco Circumcision Clamp | Mogen Circumcision Clamp | Total
Number analyzed (Participants) | 137 | 137 | 274
Age, Customized [Mean (Standard Deviation); unit: Weeks] — Gestational Age (Weeks) Population: The data of the patients who did not receive the allocated intervention were not included in the analysis.
  Weeks
    Gestational Age: number analyzed (Participants) | 121 | 130 | 251
    Gestational Age | 39.44 (1.08) | 39.29 (1.14) | 39.36 (1.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 137 | 137 | 274

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Salivary Cortisol Level
Description: Neonatal pain will be assessed by change in salivary cortisol, measured in mcg/dL., level pre and post procedure
Time Frame: Approximately 2 hours before and 15 minutes after the procedure
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Gomco Circumcision Clamp | Mogen Circumcision Clamp
Number analyzed (Participants) | 99 | 117
mcg/dL
  Pre-op Salivary Cortisol Level | 0.63 (0.59) | 0.72 (0.66)
  Post-op Salivary Cortisol Level | 1.14 (0.80) | 1.08 (0.68)

2. Primary Outcome: Post-procedure Neonatal Pain Score Using the CRIES Neonatal Pain Measurement Tool
Description: The CRIES score assigns points for crying characteristics, oxygen requirements, change in vital signs, facial expressions, and the infant's sleep state. The minimum and maximum scores of CRIES is 0 to 10, respectively with the lower score associated with lower pain and the higher score associated with high amount of pain.
Time Frame: CRIES assessment completed prior to the procedure and post procedure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Gomco Circumcision Clamp | Mogen Circumcision Clamp
Number analyzed (Participants) | 99 | 117
units on a scale | 2 [1 to 5] | 2 [0 to 6]
Statistical Analysis 1: Comparison: Gomco Circumcision Clamp vs Mogen Circumcision Clamp; Test type: Superiority or Other; p = 0.457, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the infant's hospital stay and at 4-6 weeks after discharge.
Arm/Group | Gomco Circumcision Clamp | Mogen Circumcision Clamp
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/117
Other Adverse Events (participants affected / at risk) | 0/99 | 2/117
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gomco Circumcision Clamp (N=99) | Mogen Circumcision Clamp (N=117)
Adhesion at 2 months (Surgical and medical procedures) | 0 (0) | 1 (1) — Adhesion
Pustule at head of penis - self resolved (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes